CLINICAL TRIAL: NCT07177963
Title: Cardiopulmonary Exercise Testing-based High-intensity Interval Training For Improving MAFLD
Brief Title: CPET-based HIIT for MAFLD
Acronym: CEPHIT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tang Yida (Other)
Responsible Party: Sponsor-Investigator, Tang Yida, Professor, Vice President of Peking University Third Hospital; Director of Institute of Vascular Medicine, Peking University Third Hospital; Deputy Director, State Key Laboratory of Vascular Homeostasis and Remodeling;, Peking University Third Hospital
Organization: Peking University Third Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CPHIT1
Record Dates: First submitted 2025-09-03; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Metabolic Dysfunction-Associated Fatty Liver Disease
Keywords: CPET; Exercise; HITT; Peak VO2; MAFLD
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: 54 Participants aged 35-65 years with MAFLD will be randomized 1:1 to intervention or control. The intervention group will undertake home-based HIIT four times weekly for 8 weeks. Each session comprises 8 cycles with 30-second bouts at 80% peak VO₂ followed by 60-second recoveries at 50% peak VO₂. The control group do not take any types of exercise interventions. Standard care would be provided for both groups.
Who Masked: Outcomes Assessor
Masking Description: Only blinding is maintained for data management personnel, laboratory testing personnel, and data analysts, while not applied to subjects and clinical investigators in the clinical trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIIT group (Experimental): Home-based HIIT performed on electric resistance bikes.
  Interventions: Behavioral: HIIT
- Control Group (Other): No specific exercise intervention.
  Interventions: Behavioral: No specific exercise intervention.

INTERVENTIONS:
Behavioral: HIIT — Exercise sessions were conducted as telemedically supervised, home-based HIIT performed on electric resistance bikes, with protocols individually tailored. Each HIIT session comprised 8 cycles of alternating 30-second high-intensity intervals (HIT at 80% peakVO₂) and 60-second low-intensity recovery intervals (LIT at 50% peakVO₂). Warm-up and cool-down phases were performed with the bike's resistance set to 0 watts (unloaded pedaling). The total intervention duration was 8 weeks. Received health lifestyle education based on the Prevention and Treatment Guidelines for Metabolic (Non-Alcoholic) Fatty Liver Disease (2024 Edition) and the Dietary Guidelines for Adults with Hyperlipidemia (2023 Edition).Wear smart bracelets 24/7 to monitor daily activity levels, with participants prohibited from engaging in any other systematic exercise training during the intervention period.
  Arms: HIIT group
Behavioral: No specific exercise intervention. — The control group will not receive any exercise intervention, and they will be instructed to not take any structured exercise regimens.Received health lifestyle education based on the Prevention and Treatment Guidelines for Metabolic (Non-Alcoholic) Fatty Liver Disease (2024 Edition) and the Dietary Guidelines for Adults with Hyperlipidemia (2023 Edition).Wear smart bracelets 24/7 to monitor daily activity levels, with participants prohibited from engaging in any other systematic exercise training during the intervention period.
  Arms: Control Group

SUMMARY:
High-intensity interval training (HIIT), as an individualized exercise training mode based on cardiopulmonary exercise testing (CPET), is characterized by high-intensity training sessions interspersed with short rest periods. The findings from recent trials suggest that in the management of metabolic dysfunction-associated fatty liver disease (MAFLD), compared with traditional aerobic exercise modes such as moderate-intensity continuous training, HIIT may achieve similar or even better effects in reducing liver fat content, increasing peak oxygen uptake, improving insulin resistance, and lowering blood pressure, despite requiring less time commitment and lower energy expenditure. However, there is currently no consensus regarding the formulation of HIIT exercise protocols.

Based on the lower limits of the current mainstream HIIT intensity, sets, and interval time parameters, this study aims to assess the effectiveness, safety, and feasibility of the current exercise prescription in improving MAFLD.

DETAILED DESCRIPTION:
54 Participants aged 35-65 years with MAFLD will be randomized 1:1 to intervention or control. The intervention group will undertake home-based HIIT four times weekly for 8 weeks. Each session comprises 8 cycles with 30-second bouts at 80% peak VO₂ followed by 60-second recoveries at 50% peak VO₂. The control group do not take any types of exercise interventions. Standard care would be provided for both groups.

ELIGIBILITY:
Inclusion Criteria:

Adults age 35~65 years Nonalcoholic fatty liver diagnosed by abdominal ultrasonography

In conjunction with at least one cardiometabolic risk factor:

* Overweight or Obesity: ≥ 24kg/m2，or waist circumference ≥ 90 cm in men and > 85 cm in women, or excessive body fat mass
* Prediabetes or type 2 diabetes mellitus: HbA1c ≥ 5.7%, or fasting plasma glucose ≥ 6.1mmol/L, or 2-h plasma glucose during OGTT ≥ 7.8mmol/L
* Plasma triglycerides ≥ 1.7 mmol/L (>-150 mg/dl) or lipid-lowering treatment
* HDL-cholesterol ≤ -1.0 mmol/L in men and ≤ -1.3 mmol/L in women or lipid-lowering treatment
* Blood pressure ≥ 130/85 mmHg or treatment for hypertension

Exclusion Criteria:

* Contraindications for Cardiopulmonary Exercise Testing
* The electrocardiogram (ECG) results during cardiopulmonary exercise testing (CPET) showed positive findings
* Receiving GLP-1 receptor agonists, SGLT-2i, or taking >2 antihypertensive/hypoglycemic/lipid-lowering/ antiarrhythmic drugs
* Taking dietary supplements (e.g., fish oil products, over-the-counter diet pills, meal replacements)
* Mental illness
* Other liver diseases
* Movement disorder related diseases and lower limb motor injury in the past 6 months
* Pregnant, lactating or planning to become pregnant in the near future

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-09-08 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Liver fat content (%) | Baseline (week 0) , after complete post-training (week 8).
  Liver fat content will be measured using MRI-PDFF.

SECONDARY OUTCOMES:
LSM (kPa) | Baseline (week 0) , after complete post-training (week 8).
  Liver fibrosis will be measured using MRE.
Blood specimen | Baseline (week 0) , after complete mid-training (week 4), after complete post-training (week 8).
  Lab tests include red blood cell count.
Blood specimen | Baseline (week 0) , after complete mid-training (week 4), after complete post-training (week 8).
  Lab tests include hematocrit.
Blood specimen | Baseline (week 0) , after complete mid-training (week 4), after complete post-training (week 8).
  Lab tests include hemoglobin count.
Blood specimen | Baseline (week 0) , after complete mid-training (week 4), after complete post-training (week 8).
  Lab tests include testosterone.
Blood specimen | Baseline (week 0) , after complete mid-training (week 4), after complete post-training (week 8).
  Lab tests include cortisol.
Blood specimen | Baseline (week 0) , after complete mid-training (week 4), after complete post-training (week 8).
  Lab tests include creatine kinase.
Blood specimen | Baseline (week 0) , after complete mid-training (week 4), after complete post-training (week 8).
  Lab tests include blood urea.
Blood specimen | Baseline (week 0) , after complete mid-training (week 4), after complete post-training (week 8).
  Lab tests include alanine aminotransferase.
Blood specimen | Baseline (week 0) , after complete mid-training (week 4), after complete post-training (week 8).
  Lab tests include aspartate aminotransferase.
Blood specimen | After first time and complete of mid-training (week 4), after first time and complete of post-training (week 8).
  Lab tests include lactic acid
Exercise Feasibility | Every week after complete training from week 1 to week 8.
  The implementation status of the home-based exercise prescription, including training frequency per week, average pedal frequency of the high-intensity exercise on the resistance bike, and average pedal frequency of the low-intensity exercise on the resistance bike
LSM (kPa) | Baseline (week 0) , after complete post-training (week 8).
  Liver fibrosis will be measured using Fibrotouch@.
Peak VO2 | Baseline (week 0) , after complete post-training (week 8).
  Peak VO2 is assessed through CPET, using a maximal graded treadmill test based on the Chinese expert consensus on the standardized clinical application of CPET.
BMI | Baseline (week 0) , after complete post-training (week 8).
  Weight (kg) is measured with digital weighing scale. Height (cm) is measured with a portable stadiometer. BMI is calculated as weight in kilograms divided by the square of height in meters
Brog score | After complete mid-training (week 4) , after complete post-training (week 8).
  The Borg Subjective Fatigue Scale (Borg) would be tested after each session
Exercise Feasibility | From baseline (week 0) to after complete post-training (week 8).
  The proportion of subjects leaving group during the preparation period and early termination of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Yida Tang, Study Chair — Peking University Third Hospital
Locations (5):
- China (5):
  - Beijing Ditan Hospital, Capital Medical University, Beijing
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Beijing Youan Hospital, Capital Medical University, Beijing
  - Peking University Third Hospital, Beijing
  - The Fifth Medical Center, Chinese PLA General Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No